CLINICAL TRIAL: NCT01976962
Title: Functional MR-guided Stereotactic Body Radiation Therapy of Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of adequate sample size.
Sponsor: CancerCare Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD-13-03
Record Dates: First submitted 2013-10-25; First posted 2013-11-06 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasms; Radiotherapy; Dose fractionation; Magnetic resonance imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate stereotactic body RT with MR-guided boost (Experimental): Patients will receive a dose of 36.25 Gy in 5 fractions to the entire prostate and proximal seminal vesicles with an additional boost to the dominant lesion for a total of 40 Gy in 5 fractions.
  Interventions: Radiation: Stereotactic body RT with MR-guided boost

INTERVENTIONS:
Radiation: Stereotactic body RT with MR-guided boost — Patients will receive radiotherapy over 5 fractions delivered once per week over 29 days, with 7.25 Gy per fraction to the whole prostate and 8 Gy per fraction to the dominant intraprostatic lesion. There will be a minimum of 120 hours and maximum of 192 hours between fractions. The entire course of treatment should be completed within no less than 27 days and no longer than 30 days.

SUMMARY:
To improve radiation therapy of prostate cancer, the investigators must be able to accurately identify the tumour. By using advanced functional imaging techniques available on state-of-the-art MRI scanners to clearly show the specific location of the tumour inside the prostate, the investigators can use advanced radiation therapy techniques to specifically target the tumor and control it with as few radiotherapy clinic visits as possible. This is different than current techniques which treat the whole prostate gland to the same dose, delivered over 7-8 weeks of daily radiotherapy visits. By increasing the radiation dose to the active tumor while still maintaining adequate radiation dose to the rest of the prostate, the investigators hope to better control prostate cancer and reduce complications to nearby normal tissues.

DETAILED DESCRIPTION:
This project combines advances in functional imaging of prostate cancer and hypofractionation through stereotactic body radiotherapy (SBRT), with an aim to improve tumour control and reduce or maintain normal tissue complications. The strategy will make use of the combined effectiveness of several functional imaging approaches to identify the dominant lesion(s) within the prostate. An SBRT treatment plan will be designed which utilizes 5 fractions to treat the entire prostate gland with an additional boost to the dominant lesion. The lower dose to the entire prostate should reduce normal tissue complications but still be effective in treating prostate cancer while the increased dose to the dominant lesion should improve tumour control. The use of only 5 fractions will reduce the number of patient visits, thus reducing overall treatment costs.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age >18 years
* Histologically confirmed and centrally reviewed prostate adenocarcinoma based
* PSA within 60 days
* High risk prostate cancer defined as any one of: clinical stage >= T3, Gleason score >= 8, or PSA >=20 and <50 ng/mL.

Exclusion Criteria:

* Evidence of lymph node metastasis
* Evidence of distant metastases
* Prior pelvic radiotherapy or brachytherapy
* Previous radical prostatectomy, cryotherapy, or high-frequency ultrasound
* Unable to undergo gold seed insertion
* Immunosuppressive medications
* Inflammatory bowel disease
* Unable to undergo MRI
* Previous bilateral orchiectomy
* Previous hormonal therapy including LHRH agonists (leuprolide, goserelin), LHRH antagonists (degarelix), anti-androgens (bicalutamide, flutamide, nilutamide), surgical castration, and estrogens
* Previous finasteride within 14 days.
* Previous dutasteride within 180 days.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Quality of Life as per EPIC | 6 months
  Expanded Prostate Cancer Index Composite (EPIC) bowel domain

SECONDARY OUTCOMES:
Quality of Life as per EPIC and SF-12 | Up to 5 years
  Expanded Prostate Cancer Index Composite (EPIC) questionnaire (other domains) and Medical Outcomes Study Short-Form 12 (SF-12) v2
GU and GI Toxicity | Up to 5 years
  RTOG and CTCAE v4.0 genitourinary and gastrointestinal toxicities
Biochemical failure | 5 years
  Phoenix defined (nadir PSA + 2 ng/mL) biochemical failure
Pathologic response | 3 years
  Pathologic presence of malignancy on biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Aldrich Ong, MD, Principal Investigator — CancerCare Manitoba
Locations (1):
- CancerCare Manitoba, Winnipeg, Manitoba, Canada